CLINICAL TRIAL: NCT02454621
Title: Randomized Controlled Trial of the Smoking Cessation Volitional Help Sheet in Primary Care
Brief Title: Trial of the Smoking Cessation Volitional Help Sheet in Primary Care
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The researcher quit the study
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Christopher Armitage, Professor of Health Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAN-CA-01
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Participants read a brief statement designed to encourage them to quit smoking ("We want you to plan to quit smoking"). Participants are presented with a table with two columns and twenty rows. Twenty critical situations (temptations) are presented in the left hand column and 20 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to smoke and identifying ways to overcome those temptations had been shown to promote smoking cessation and are asked to tick critical situations/appropriate responses that might be useful to them.
  Interventions: Behavioral: Volitional help sheet
- Volitional help sheet (Experimental): Participants read a brief statement designed to encourage them to quit smoking ("We want you to plan to quit smoking"). Participants are presented with a table with two columns and twenty rows. Twenty critical situations (temptations) are presented in the left hand column and 20 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to smoke and identifying ways to overcome those temptations had been shown to promote smoking cessation. Implementation intentions are formed by linking critical situations with appropriate responses by drawing lines between critical situations and appropriate responses.
  Interventions: Behavioral: Volitional help sheet

INTERVENTIONS:
Behavioral: Volitional help sheet — Participants are asked to form implementation intentions using a volitional help sheet (Armitage, 2008).

SUMMARY:
The study will recruit patients who smoke from a general practice clinic and randomize them either to: (1) form implementation intentions by linking in memory situations in which they are tempted to smoke with strategies to avoid smoking in those situations using a volitional help sheet, or (2) to consider the situations in which they are tempted to smoke alongside possible strategies to avoid smoking as presented in the volitional help sheet but not to form implementation intentions. The effects on self-reported smoking will be assessed 1 month post-intervention.

DETAILED DESCRIPTION:
The study will recruit patients who smoke from a general practice clinic and randomize them either to: (1) form implementation intentions by linking in memory situations in which they are tempted to smoke with strategies to avoid smoking in those situations using a volitional help sheet, or (2) to consider the situations in which they are tempted to smoke alongside possible strategies to avoid smoking as presented in the volitional help sheet but not to form implementation intentions. The effects on self-reported smoking will be assessed 1 month post-intervention.

Design: This study will use questionnaires to assess participants smoking habits and then employ planning strategies to help then quit. Follow up questionnaires will be used to ascertain the success of planning on smoking cessation.

Sample Size: Upon entry to the General Practice (GP) clinic participants will be made aware of the study by the receptionist and asked to complete a copy if they are a smoker. The investigators are looking to recruit a minimum of fifty participants for each condition, but aim to collect data from as many participants as possible during the recruitment phase.

Recruitment: To participate in this study a person must be over the age of 18 and a smoker. The receptionists at the GP clinic will inform people of the study on entry and ask that they complete the questionnaire should they be 18 (or older) and smoke.

Procedure: Participants will be recruited from a GP clinic in Birmingham. They will be asked by the receptionists, upon entry to the clinic, to take one of the investigators' questionnaire packs if they are a smoker. These packs will be displayed on a table beside the reception desk. The packs begins with a briefing sheet that provides information about both how to complete the questionnaire and the reason for the study. The sheet will also inform participants that they do not have to complete the questionnaire that day, and they should feel free to come back and take part at a later date. It will also indicate to participants that they can withdraw from the study at any time, and a reason does not need to be provided. Once they have read the briefing sheet and generated their personal identity code, as instructed, they will complete the questionnaire. Completed questionnaires will be returned to the returns box. This will be securely stored in the GP clinic and collected once a week. Data from all packs will be collected and transferred to a secure university server before being shredded. A month after the participants have completed the initial questionnaire they will receive a follow-up questionnaire; either via e-mail or a hard copy via post where indicated. Data from the online questionnaire will be collected immediately, hard copy questionnaires will be returned via a pre-paid envelope (enclosed with the hard copy questionnaire) and transcribed onto a secure university computer before being shredded. Participants contact information will be kept separate from the data. Once participants have completed the follow-up questionnaire their involvement in the study is over.

Outcomes and Analysis: The main purpose of this study is to explore the role of planning in encouraging people to quit smoking when recruited by receptionists in a GP clinic. Quantitative analysis will be conducted to assess the effects of planning on smoking cessation. The investigators expect to find that planning is effective in helping people quit, and that the questionnaire is compatible for use within a healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* smoker

Exclusion Criteria:

* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Quitting smoking | 1 month
  Self-reported smoking cessation
Nicotine dependence | 1 month
  Self-reported nicotine dependence

SECONDARY OUTCOMES:
Habit | 1 month
  Self-reported habit (e.g., "Smoking is something I do automatically: strongly disagree-strongly agree")
Action control | 1 month
  Self-reported action control (e.g., "During the last week I often had my intention to quit smoking on my mind: strongly disagree-strongly agree")
Craving | 1 month
  Self-reported craving
Self-identity | 1 month
  Self-reported self-identity (e.g., "Smoking is an important part of who I am: strongly disagree-strongly agree")

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Armitage, PhD, Principal Investigator — University of Manchester
Locations (1):
- Sandwell and West Birmingham CCG, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Result] Armitage CJ. A volitional help sheet to encourage smoking cessation: a randomized exploratory trial. Health Psychol. 2008 Sep;27(5):557-66. doi: 10.1037/0278-6133.27.5.557. PMID 18823182